CLINICAL TRIAL: NCT06225531
Title: Exploring the Feasibility and Acceptability of an Autobiographical Memory-Based Intervention for People With Suicidality: A Case Series
Brief Title: An Autobiographical Memory-Based Intervention for Suicidality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Alexandra Powell, Trainee Clinical Psychologist, Lancaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 316697
Record Dates: First submitted 2024-01-05; First posted 2024-01-26 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Suicidal Ideation; Mental Health Disorder
Keywords: Suicide; Autobiographical Memory
MeSH Terms: conditions — Suicidal Ideation; Mental Disorders; Suicide

STUDY DESIGN:
Intervention Model Description: Experimental case series, with a non-concurrent multiple baseline design. This will involve a baseline period which varies in length between participants (3-5 sessions), followed by an intervention period (6 sessions for all)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autobiographical Memory Based Intervention (Experimental): All participants will be placed into the intervention arm, in which the participants will receive 6 autobiographical memory based intervention sessions, lasting approximately one hour.
  Baseline lengths will vary from 3 - 5 sessions, with the initial session lasting approximately one hour, and follow up sessions lasting approximately 30 minutes. This randomisation is 1) to enable the effects of treatment to be separated from the effects of time seen clinically and 2) in order to control for the therapeutic value of contact.
  Interventions: Other: Autobiographical Memory Based Intervention

INTERVENTIONS:
Other: Autobiographical Memory Based Intervention — The intervention involves 6 sessions of therapeutic input based around autobiographical memories. Memory based activities will broadly follow the 5 stages outlines in the broad-minded affective coping (BMAC) procedure, but with a focus on specific memories. It will follow the following structure:
  Session 1 - Introduction and Familiarisation Session 2 - Neutral Memories Session 3 - Positive Memories Session 4 - Memories of Moves Away from Suicidality Session 5 - Practice of Preferred Memory (from Sessions 2-4) Session 6 - Continued Practice and Post-Intervention Planning

SUMMARY:
The study involves a short therapy intervention for people who are experiencing thoughts of suicide. The intervention will focus upon different memories from the person's life. These memories will vary in the emotions they evoke - some memories will be associated with neutral emotions, whereas others will bring up positive emotions. The intervention will have a particular focus upon memories of times when the participants have moved away from thinking about suicide, with the aim of reinforcing memories of what helped them to reconnect with life. The intervention will also introduce relaxation techniques, in addition to involving a safety planning component. The project aims to consider whether this intervention is acceptable and feasible for this population.

DETAILED DESCRIPTION:
This study is looking at whether an autobiographical memory-based intervention is acceptable and suitable for people with thoughts of suicide within a secondary mental health population. Autobiographical memory involves the recollection of past events in a person's own life, and this has been linked to a person's sense of identity, goals, and orientation in the present. Memories linked to negative emotions have been shown to be durable, accessible, and easily and vividly remembered. The power that memories of suicidal ideation and suicide attempts hold is therefore concerning. This intervention aims to support participants to more readily access positive and neutral autobiographical memories, using memory tasks and worksheets. By focusing upon individuals' moves away from suicidal thinking, it also aims to shift the focus onto remembering what led people to reconnect with life.

The study is an experimental case series using a non-concurrent A-B multiple baseline design, in which the participants first attend 3-5 baseline sessions prior to attending 6 intervention sessions. Sessions are one-to-one. The initial baseline session and all intervention sessions will take place face-to-face. The follow-up baseline sessions can be conducted in-person, online via Microsoft Teams, or via telephone, depending on participant preference.

The initial baseline session will involve assessing risk and updating participants' safety plan. The intervention involves 6 sessions of approximately one hour. The first session will focus upon familiarisation to concepts in the intervention, using imagery-based metaphors to support understanding. Sessions 2-4 will focus on different memories - neutral, positive, and memories of moves away from suicidal thinking. Memory tasks will broadly follow the 5 stages outlined in the broad-minded affective coping (BMAC) procedure, but with a focus on these specific memories. In the final 2 sessions, participants will have a choice around which memory to focus on. The final session will also involve post-intervention planning. Outcome measures will be completed in all baseline and intervention sessions.

The study aims to recruit 5-7 participants from community mental health teams (CMHTs) in which supervisory support can be arranged. The intervention will be conducted by the principle investigator (AP), a trainee psychologist, under the supervision of clinical psychologists within the CMHTs (JK and NI) who are also members of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Individual has experienced suicidal ideation and/or suicidal behaviours within the previous 3 months. This will be screened for by asking the questions:

  1. Have you had thoughts or images of ending your life within the past three months? or
  2. Have you attempted to end your life within the past 3 months?
* Currently under a Community Mental Health Team (CMHT) within which supervisory support can be arranged.

Exclusion Criteria:

* Moderate/severe learning disability
* Organic cerebral disease/injury which significantly affects language comprehension or expression
* Non-English speaking
* Acute psychosis which would affect engagement
* Receiving psychological treatment or participating in another research intervention
* At imminent risk of acting upon thoughts of suicide or of harm to others. This will be screened for by assessing for the presence of active intent or plans to harm themselves or others within the next month. If these individuals consent to be contacted again after a month, the researcher will consider approaching them again to assess for changes to imminent risk. If the individual met the eligibility criteria at this point, the individual would be invited to take part in the study.
* A history of violence or harm to others to a degree in which clinicians have assessed one-to-one sessions to be unsafe
* Currently within an inpatient setting or open to a home-based treatment team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Acceptability - Therapeutic Alliance | Up to 14 weeks
  This is to consider the therapeutic relationship between the practitioner and participant. Measured using the Working Alliance Inventory - Short Revised, scored out of 60 where a high score indicates strong alliance.
Acceptability - Adverse effects | Up to 14 weeks
  This is to assess for any negative outcomes of the intervention. Measured using the Adverse Effects in Psychotherapy questionnaire, with statements scored on a 5 point scale from 'not at all' to 'very much'
Acceptability - Clinical Global Impression | Up to 14 weeks
  This is a measure of the practitioner's overall clinical impression of the participant during the session. This is measured using the Clinical Global Impressions Scale, where severity is scored on a scale of 1-7 (where 7 indicates a negative impression/change).
Acceptability - Overall | Up to 14 weeks
  The overall acceptability of the intervention will be measured using an adapted Acceptability Scale. This includes measures of multiple key areas which are important for an intervention to be classified as acceptable by a participant. Statements are assessed on a 5 point scale from 'strongly disagree' to 'strongly agree'.
Acceptability - Qualitative Feedback | Up to 14 weeks
  Qualitative feedback around the acceptability of the intervention - collected at the end of the Adverse Effects in Psychotherapy Scale with the question 'If you would like to describe your experience of taking part in the study in your own words, please use the following space'.
Feasibility - rates of recruitment, attendance, and completion | Up to 14 weeks
  To assess whether the intervention is feasible within this population, the investigators will consider the proportion of participants approached who met the eligibility criteria, and proportion of these who consent to taking part in the study. The investigators will also collect data on attendance rates, where reasonable attendance will be set as ≥ 3 sessions out of the 6-session intervention, in accordance with the criteria set out in a similar case series study. Therapy completion rates will also be recorded, where the investigators will look at the number of participants who completed the final set of therapy measures.

SECONDARY OUTCOMES:
Suicidality | Up to 14 weeks
  Measured using the Columbia Suicide Severity Rating Scale. The scale uses yes/no questions, plus an overall score of actual lethality (where 0 is least severe and 5 is most) and of potential severity (where 0 is lowest risk and 2 is highest risk) in relation to the individual's i) most recent suicide attempt, ii) most lethal attempt, and iii) first attempt.
Entrapment | Up to 14 weeks
  Entrapment has been closely linked to suicidal ideation and suicide risk. The investigators will measure this using a 4-item Entrapment Scale - Short-Form. This is scored out of 16, where a high score indicates high levels of entrapment.
Perceived Burdensomeness / Thwarted Belonging | Up to 14 weeks
  Interpersonal factors have also been linked to suicidal ideation and suicide risk. This will be measured using the Interpersonal Needs Questionnaire. This is scored out of 105, where a high score indicates greater levels of perceived burdensomeness and thwarted belonging.

OTHER OUTCOMES:
Sessional Mood Scale | Up to 14 weeks
  Participants' mood from 1-10 will be rated at the start of each session to assess for weekly changes, where 10 indicates the most positive mood.

CONTACTS AND LOCATIONS:
Overall Officials: James Kelly, ClinPsyD, Principal Investigator — Lancaster University
Locations (1):
- Greater Manchester Mental Health NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gershman SJ. Predicting the Past, Remembering the Future. Curr Opin Behav Sci. 2017 Oct;17:7-13. doi: 10.1016/j.cobeha.2017.05.025. Epub 2017 Jun 9. PMID 28920071
- [Background] Johnson, J., Gooding, P.A., Wood, A.M. et al. A Therapeutic Tool for Boosting Mood: The Broad-Minded Affective Coping Procedure (BMAC). Cogn Ther Res 37, 61-70 (2013). https://doi.org/10.1007/s10608-012-9453-8
- [Background] Hatcher, R. L., & Gillaspy, J. A. (2006). Development and validation of a revised short version of the working alliance inventory. Psychotherapy Research, 16(1), 12-25. https://doi.org/10.1080/10503300500352500
- [Background] Hutton, P. (2016). Positive Clinical Psychology and the Promotion of Happiness, Compassion, and Autonomy in People with Psychosis. In The Wiley Handbook of Positive Clinical Psychology (pp. 245-260). https://doi.org/https://doi.org/10.1002/9781118468197.ch17
- [Background] Gilbert P, Allan S. The role of defeat and entrapment (arrested flight) in depression: an exploration of an evolutionary view. Psychol Med. 1998 May;28(3):585-98. doi: 10.1017/s0033291798006710. PMID 9626715
- [Background] De Beurs D, Cleare S, Wetherall K, Eschle-Byrne S, Ferguson E, B O'Connor D, C O'Connor R. Entrapment and suicide risk: The development of the 4-item Entrapment Scale Short-Form (E-SF). Psychiatry Res. 2020 Feb;284:112765. doi: 10.1016/j.psychres.2020.112765. Epub 2020 Jan 9. PMID 31945600
- [Background] Talmi D, Anderson AK, Riggs L, Caplan JB, Moscovitch M. Immediate memory consequences of the effect of emotion on attention to pictures. Learn Mem. 2008 Mar 5;15(3):172-82. doi: 10.1101/lm.722908. Print 2008 Mar. PMID 18323572
- [Background] Williams JM, Barnhofer T, Crane C, Herman D, Raes F, Watkins E, Dalgleish T. Autobiographical memory specificity and emotional disorder. Psychol Bull. 2007 Jan;133(1):122-48. doi: 10.1037/0033-2909.133.1.122. PMID 17201573
- [Background] Williams SE, Ford JH, Kensinger EA. The power of negative and positive episodic memories. Cogn Affect Behav Neurosci. 2022 Oct;22(5):869-903. doi: 10.3758/s13415-022-01013-z. Epub 2022 Jun 14. PMID 35701665
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Taylor CDJ, Bee PE, Kelly J, Emsley R, Haddock G. iMAgery focused psychological therapy for persecutory delusions in PSychosis (iMAPS): a multiple baseline experimental case series. Behav Cogn Psychother. 2020 Sep;48(5):530-545. doi: 10.1017/S1352465820000168. Epub 2020 Apr 8. PMID 32264985
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671